CLINICAL TRIAL: NCT06519903
Title: The Impact of Breathing Exercises on Anxiety Levels During the First Insulin Injection in Patients With Type 2 Diabetes-the BREATH Study
Brief Title: Anxiety Reduction in Type 2 Diabetes Through Breathing ExercisesPatients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Goztepe Prof Dr Suleyman Yalcın City Hospital (Other)
Responsible Party: Principal Investigator, Ayse N Erbakan, Principal Investigator, Goztepe Prof Dr Suleyman Yalcın City Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Breath Study
Record Dates: First submitted 2024-07-14; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Type 2 Diabetes; Type 2 Diabetes Treated With Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BREATH Intervention Group (Active Comparator): During initial meeting before randomization, all patients was administered the SUDS, STAI-I, and STAI-II scales by another clinical nurse. Following this, patients were taken to a quiet, well-ventilated, and well-lit room for the BREATH breathing technique session. Following a brief training session, the BREATH technique was applied in individual sessions lasting approximately 24 min. The post-test SUDS, STAI-I, and STAI-II scales were administered by the clinical nurse.
  Interventions: Behavioral: BREATH technique
- Control Group (No Intervention): Patients in the control group were administered the Demographic Information Form, SUD, STAI-I, and STAI-II as a pre-test. No intervention was administered in the control group. After the pre-test, the patient was placed in a quiet, well-ventilated, and well-lit room for 24 minutes. Subsequently, the SUD, STAI-I, and STAI-II scales were administered as post-tests.

INTERVENTIONS:
Behavioral: BREATH technique — The BREATH techniques include deep breathing, rapid breathing, and alternate nostril breathing exercises. Participants were first instructed on the breathing exercises (at the lowest point of breathing, close the left nostril with the right index finger and exhale through the right nostril): Breathe in through the right nostril, then close it with your thumb and breathe out through the left nostril. This cycle was repeated at least three more times.
  Arms: BREATH Intervention Group

SUMMARY:
Injection-related anxiety is a significant barrier to the management of type 2 diabetes, adversely affecting treatment adherence and glycemic control. This study investigated the effectiveness of breathing exercises in reducing anxiety during the first insulin injection.

DETAILED DESCRIPTION:
This study is designed as a randomized, double-blind, experimental study. Data from patients who agree to participate in the study was collected by the researcher prior to testing. Variables collected include age, gender, marital status, education level, occupation, body mass index (BMI), HbA1c levels and diabetes duration, as well as scores on the Subjective Disorders Scale (SUDS), State Anxiety Inventory (STAI-I) and Trait Anxiety Inventory (STAI-II). Patients were then randomly assigned to the intervention (BREATH) and control groups using a computer-generated randomization table. Allocation continued until the blocks in each group are equal in size.

Participants in the BREATH and control groups was identified prior to the intervention. All participants completed a form with demographic information. The participants in the control group completed the SUDS, STAI-I and Trait Anxiety Inventory (STAI-II) scales before the test. They then had 30 minutes of free time. The SUDS, STAI-I and STAI-II scales were then completed for the post-test.

In the BREATH intervention group, participants were first instructed on the breathing exercises (at the lowest point of breathing, close the left nostril with the right index finger and exhale through the right nostril). Breathe in through the right nostril, then close it with your thumb and breathe out through the left nostril. This cycle was repeated at least three more times. Participants completed the SUDS, STAI-I and STAI-II scales before the test, following by a single BREATH session (approximately 30 minutes). After the test, the SUDS, STAI-I and STAI-II were administered.

Standard treatment for all patients was not interrupted during the study. Appointments for the randomized patients were made by telephone to avoid encounters and mutual interference between the groups.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes diagnosis for at least one year,
* followed up at the diabetes outpatient clinic,
* literate and able to understand and complete study forms,
* first-time insulin injectors in addition to oral antidiabetics,

Exclusion Criteria:

* younger than 18 years
* older than 65 years
* having visual, auditory, or mental impairments that would affect to complete the forms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
the impact of breathing exercises on anxiety levels during the first insulin injection in patients with type 2 diabetes, the evaluation of distress | thirty minutes
  Anxiety levels were determined by Subjective Units of Disturbance Scale test. The Subjective Units of Disturbance Scale (SUDS) is a self-report measure developed by Joseph Wolpe to quantify an individual's level of distress. The scale ranges from 0 to 10, where
  * 0 represents no distress or disturbance.
  * 10 represents the highest level of imaginable distress or disturbance.
the impact of breathing exercises on anxiety levels during the first insulin injection in patients with type 2 diabetes, the evaluation of current anxiety | thirty minutes
  Anxiety levels were determined by State Anxiety Inventory tests The State Anxiety Inventory is a widely used self-report questionnaire designed to assess the current state of anxiety, distinguishing it from trait anxiety (which is more about general anxiety tendencies). The total score ranges from 20 to 80, with higher scores indicating higher state anxiety levels.
the impact of breathing exercises on anxiety levels during the first insulin injection in patients with type 2 diabetes, the evaluation of axiety state | thirty minutes
  The Trait Anxiety Inventory is part of the State-Trait Anxiety Inventory and specifically measures trait anxiety, which refers to relatively stable individual differences in anxiety proneness and the tendency to perceive stressful situations as threatening.The total score ranges from 20 to 80, with higher scores indicating higher trait anxiety levels.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse N Erbakan, Principal Investigator — Istanbul Goztepe Prof. Dr. Suleyman Yalcin City Hospital
Locations (1):
- SB Istanbul Goztepe Prof Dr Suleyman Yalcin City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No